CLINICAL TRIAL: NCT06582654
Title: URINORM: Normalizing Antibody Detection in First-void Urine
Brief Title: Normalizing Antibody Detection in First-void Urine
Acronym: URINORM
Status: Recruiting | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Wiebren Tjalma, Professor and Gynecological Oncologist, Universiteit Antwerpen
Other Study IDs: B3002023000105
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Human Papillomavirus Infection
Keywords: Antibodies; Vaccination; Self-sampling; First-void urine
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — First-void urine samples Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Pre-adolescent group: Defined as girls between 9 and 14 years old, who are vaccinated against HPV with either the Cervarix, Gardasil or Gardasil9 vaccine and are not yet menstruating (pre-menarche).
  Interventions: Device: Sampling
- Ovulatory group: Defined as women between 18 and 30 years old, who are vaccinated against HPV with either the Cervarix, Gardasil or Gardasil9 vaccine and are not using any hormone- or ovulation-influencing contraceptives that impact hormonal levels during the menstrual cycle.
  Interventions: Device: Sampling
- Ovulation-influencing contraceptive group: Defined as women between 18 and 30 years old, who are vaccinated against HPV with either the Cervarix, Gardasil or Gardasil9 vaccine and are using ovulation-influencing contraceptives that impact hormonal levels during the menstrual cycle (including oral contraceptives, hormonal ring, contraceptive injection, contraceptive patch, hormonal implant).
  Interventions: Device: Sampling
- Non-ovulation-influencing contraceptive group: Defined as women between 18 and 30 years old, who are vaccinated against HPV with either the Cervarix, Gardasil or Gardasil9 vaccine and are using contraceptives that do not affect ovulation (i.e. intrauterine devices).
  Interventions: Device: Sampling
- Post-menopausal group: Defined as fully vaccinated women between 50 and 70 years old, who are vaccinated against HPV with either the Cervarix, Gardasil or Gardasil9 vaccine and have had no menses for at least one year.
  Interventions: Device: Sampling
- Male group: Defined as fully vaccinated men between 18 and 30 years old, who are vaccinated against HPV with either the Cervarix, Gardasil or Gardasil9 vaccine.
  Interventions: Device: Sampling

INTERVENTIONS:
Device: Sampling — Collection of first-void urine (i.e. the initial stream of the urine) with the Colli-Pee device (Novosanis, Belgium) (6-21 samples over a period of 36 days).
  Collection of blood samples (2 samples, at day 1 and 36 of the study).

SUMMARY:
The aim of this study is to develop robust analytical protocols for the monitoring of vaccine induced immunity against the Human Papillomavirus (HPV) in first-void urine samples and to examine fluctuations of urinary HPV-specific antibodies and potential normalization markers in different cohorts.

DETAILED DESCRIPTION:
To date, invasive clinician-collected cervical samples, blood, and vaginal samples are still the primary methods to monitor disease and immune responses to vaccine-preventable genital tract infections. Replacing these samples with a specimen that is non-invasive and can be self-collected at home could have important acceptance and feasibility advantages and could facilitate the logistics of clinical trials and future epidemiological studies. Initial results of experiments using first-void urine samples for immune response monitoring are promising. However, overall standardization and normalization of fluctuation in signals are necessary for it to become a suitable genital tract liquid biopsy in vaccine research. Therefore, the aim of this study is to normalize antibody detection in first-void urine by reducing sample variability, using the human papillomavirus (HPV) as a model.

A total of 150 participants will be included, consisting of six different cohorts, including a group of pre-adolescent girls (n=25), a group of young women using ovulation-influencing contraceptives (n=25), a group of young women using non-ovulation-influencing contraceptives (n=25), a group of young women using no contraceptives (n=25), a group of post-menopausal women (n=25), and a group of men (n=25). Participants will be followed over a period of 36 days, and will be asked to self-collect 6 to 21 first-void urine samples (depending on cohort) using a Colli-Pee 20mL (Novosanis). Moreover, participants will have two scheduled visits (day 1 and 36 of the study) at the study site, where each time a blood collection (1x 5-10cc) will be performed.

Collected first-void urine and serum samples will be analyzed for menstrual cycle-related fluctuations and between-group differences in HPV-specific antibody levels. Moreover, to compare immunological with viral endpoints, HPV DNA detection and genotyping will be performed on the first-void urine sample and samples will be tested for various biomarkers that might be valuable for the normalization of inter- and intra-individual variability.

ELIGIBILITY:
Inclusion Criteria:

* Vaccinated with either the Cervarix, Gardasil or Gardasil9 HPV-vaccine and able to present vaccination booklet or another official document proving this.
* Able to understand the information brochure and what the study is about.
* Willing to give informed consent to contact his/her general practitioner and/or gynecologist to access details on their HPV vaccination schedule and, in case a woman within the screening population, cervical cancer screening results (smears, HPV tests, colposcopy, biopsy).

Exclusion Criteria:

* Participating in another clinical trial at the same time of participating in this study.
* Women that underwent hysterectomy or were treated for cervical (pre)cancer lesions within the six months prior to study enrolment.
* Pregnant women.
* Being positive for Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C.
* Having a history or current evidence of any condition or abnormality that might confound the results of the study or is not in the best interest of the individual to participate, in the opinion of the investigator.

Ages: 9 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — All groups are female, except for one male group (aged 18-30 years old)
Study Population: A total of 150 participants will be included, consisting of six different cohorts, including a group of pre-adolescent girls (n=25), a group of young women using ovulation-influencing contraceptives (n=25), a group of young women using non-ovulation-influencing contraceptives (n=25), a group of young women using no contraceptives (n=25), a group of post-menopausal women (n=25), and a group of men (n=25).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of total and HPV-specific IgG (immunoglobulin G) in first-void urine. | Within six months after completion of the study
  To follow-up levels of total and HPV-specific antibodies in first-void urine at repeated measurements and compare levels of total and HPV-specific antibodies in first-void urine between young men, pre-adolescent girls, post-menopausal women, and women on a contraceptive or ovulatory cycle.

SECONDARY OUTCOMES:
Concentration of total and HPV-specific IgG (immunoglobulin G) in serum. | Within six months after completion of the study
  To compare levels of total and HPV-specific antibodies in serum at repeated measurements and look into correlation between total and HPV-specific antibodies in serum and first-void urine.
HPV DNA status of first-void urine samples. | Within six months after completion of the study
  To test for the presence of HPV DNA in first-void urine samples from different cohorts of men, girls and women vaccinated against HPV.
Other biomarkers/analyses. | Within six months after completion of the study
  To test various biomarkers (e.g. total IgG, IgG subclasses, total protein, total human DNA…) in first-void urine samples from different cohorts of men, girls and women vaccinated against HPV and perform other relevant analyses within the scope of the study.
  To test various biomarkers (e.g. total IgG, IgG subclasses, total protein, total human DNA…) in first-void urine samples from different cohorts of men, girls and women vaccinated against HPV and perform other relevant analyses within the scope of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Wiebren Tjalma, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University of Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No